CLINICAL TRIAL: NCT00000264
Title: Subjective/Psychomotor/ Effects of Combined Alcohol & Nitrous Oxide
Brief Title: Subjective/Psychomotor/ Effects of Combined Alcohol & Nitrous Oxide - 16
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Model: Crossover | Masking: Double
Other Study IDs: NIDA-08391-16; R01DA008391 (NIH); R01-08391-16
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; inhalant; ethanol; subjective effects; psychomotor effects; healthy volunteer
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Nitrous Oxide; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- 0 g/Kg ethanol +/- 30% nitrous oxide (Placebo Comparator)
  Interventions: Drug: 30% Nitrous oxide; Other: 0 g/Kg ethanol
- 0.35 g/Kg ethanol +/- 30% nitrous oxide (Active Comparator)
  Interventions: Drug: 30% Nitrous oxide; Other: 0.35 g/Kg ethanol
- 0.7 g/Kg ethanol +/- 30% nitrous oxide (Active Comparator)
  Interventions: Drug: 30% Nitrous oxide; Other: 0.7 g/Kg ethanol

INTERVENTIONS:
Drug: 30% Nitrous oxide
Other: 0.35 g/Kg ethanol
  Arms: 0.35 g/Kg ethanol +/- 30% nitrous oxide
Other: 0.7 g/Kg ethanol
  Arms: 0.7 g/Kg ethanol +/- 30% nitrous oxide
Other: 0 g/Kg ethanol
  Arms: 0 g/Kg ethanol +/- 30% nitrous oxide

SUMMARY:
The purpose of this study is to examine the subjective, psychomotor, and reinforcing effects of combined alcohol and nitrous oxide intake in healthy volunteers.

ELIGIBILITY:
Please contact site for information.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 1997-09; Primary Completion 1999-10 (Actual); Study Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
Mood | Baseline and post inhalation
Psychomotor performance | Baseline and post inhalation
Cognitive performance | Baseline and post inhalation
Choice of nitrous oxide vs placebo | after each ethanol session

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States